CLINICAL TRIAL: NCT07115368
Title: An Umbrella Phase 1b, Open-label, Multi-Cohort Study to Evaluate Safety, Pharmacokinetics, and Antiviral Activity of Novel Antiretrovirals in Participants With HIV-1; Substudy-04: GS-1219
Brief Title: Study of GS-1219 in Participants With HIV-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate study.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-544-5905-04
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 of GS-1219 (Experimental): Participants in Cohort 1 will receive a single dose of GS-1219 800 mg administered once daily on Day 1 through Day 4, followed by a single dose of GS-1219 800 mg administered on Day 7, all in the fasted condition.
  After assessments on Day 11 or upon early termination (ET), the participants initiate a regimen of bictegravir/emtricitabine/tenofovir alafenamide (Biktarvy®) (BVY), or an alternative standard of care (SOC) antiretroviral (ART) regimen (example INSTI + NRTIs: dolutegravir (DTG)/abacavir (ABC)/3TC or DTG/3TC) up to Day 25.
  Following the completion of Cohort 1, additional cohorts may open for enrollment if further data are needed. Participants will receive single or multiple doses of GS-1219 up to 1800 mg administered in the fasted condition or with food (low-fat or high-fat meal).
  Interventions: Drug: GS-1219; Drug: BVY; Drug: Standard of Care

INTERVENTIONS:
Drug: GS-1219 — Administered orally
Drug: BVY — Administered orally
  Other Names: Biktarvy®
Drug: Standard of Care — Antiretroviral therapy, administered orally non nonnucleoside reverse transcriptase inhibitor (NNRTIs), examples: ABC/ DTG/3TC; DTG plus (TAF or TDF) plus (FTC or 3TC)

SUMMARY:
This study is part of a master study. The goal of master protocol (GSUS-544-5905, NCT05585307) is to learn how novel antiretrovirals (medicines that stop the virus from multiplying) affect the human immunodeficiency virus-1 (HIV-1) infection in people living with HIV (PWH).

Substudy GS-US-544-5905-04 is to learn more about study drug GS-1219, safety, pharmacokinetics (PK) (how GS-1219 is absorbed, modified, distributed, and removed from the body of the participants), and antiviral activity in Participants With HIV-1.

DETAILED DESCRIPTION:
To refer master study protocol (GS-US-544-5905), refer to NCT05585307 on https://clinicaltrials.gov/

ELIGIBILITY:
Key Inclusion Criteria:

All Substudies:

* Plasma human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) ≥ 5000 copies/mL but ≤ 400,000 copies/mL at screening.
* Cluster of differentiation 4 (CD4) cell count > 200 cells/mm^3 at screening.
* Antiretroviral (ARV) treatment-naive or treatment-experienced but naive to the investigational ARV drug class being investigated in the given substudy and have not received any ARV within 12 weeks of screening, including medications received for pre-exposure prophylaxis (PrEP) or postexposure prophylaxis (PEP) (note that current or prior receipt of long acting (LA) parenteral ARVs such as monoclonal antibodies (mAbs) targeting HIV-1, injectable cabotegravir (CAB), injectable rilpivirine (RPV) or injectable Lenacapavir (LEN) is exclusionary).
* Have adequate renal function (estimated glomerular filtration rate (eGFR) ≥ 70 mL/min/1.73 m^2)
* No clinically significant abnormalities in electrocardiogram (ECG) at screening.

Substudy-04:

* Willing to initiate BVY provided by the sponsor, or an alternative SOC ART regimen selected by the investigator on Day 11 or upon ET.
* Willing and able to comply with meal requirements on dosing days.

Key Exclusion Criteria:

* Known historical genotypic or phenotypic resistance to 4 major ARV classes (nucleoside reverse transcriptase inhibitor (NRTI), nonnucleoside reverse transcriptase inhibitor (NNRTI), protease inhibitor (PI), integrase strand-transfer inhibitor (INSTI)).
* History of an AIDS-defining condition including present at the time of screening.
* Active, serious infections (other than HIV-1) requiring therapy and including active tuberculosis infection < 30 days prior to randomization.
* History of or current clinical decompensated liver cirrhosis (eg, ascites, encephalopathy, or variceal bleeding).
* Any other serious or active clinical condition or prior therapy that, in the opinion of the investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements.
* Hepatitis C virus (HCV) antibody positive and detectable HCV RNA.
* Chronic hepatitis B virus (HBV) infection, as determined by either:

  1. Positive HBV surface antigen and negative HBV surface antibody, regardless of HBV core antibody status, at the screening visit, or
  2. Positive HBV core antibody and negative HBV surface antibody, regardless of HBV surface antigen status, at the screening visit.
* Hepatic transaminases (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) > 5 x upper limit of normal (ULN).
* Current alcohol or substance use judged by the investigator to potentially interfere with individual study compliance.
* Positive serum pregnancy test at screening or a positive pregnancy test prior to Day 1.
* Individuals with plan to breastfeed during the study period including the protocol-defined follow-up period.
* Requirement for ongoing therapy with or prior use of any prohibited medications listed in the protocol. Any prescription medications or over the counter medications, including herbal products, within 28 days prior to start of study drug dosing must be reviewed and approved by the sponsor, with the exception of vitamins and/or acetaminophen and/or ibuprofen.
* Any current or prior receipt of LA parenteral ARVs such as mAbs targeting HIV-1, injectable CAB, or injectable RPV, or injectable LEN, for treatment or prophylaxis (PrEP, PEP).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-08-11 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Plasma Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) (log10 Copies/mL) at Day 11 Relative to Historical Placebo Data | Baseline, Day 11

SECONDARY OUTCOMES:
Change From Baseline in Plasma HIV-1 RNA (log10 Copies/mL) at Day 8 Relative to Historical Placebo Data | Baseline, Day 8
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) | First dose up to Day 25
Percentage of Participants With Graded Laboratory Abnormalities | First dose up to Day 25
Pharmacokinetic (PK) Parameter: Cmax of GS-1219 | Day 1 Predose up to Day 11
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: AUC of GS-1219 | Day 1 Predose up to Day 11
  AUC is defined as the area under the concentration versus time curve (AUC).
PK Parameter: Ct of GS-1219 | Any day between Day 1 Predose up to Day 11
  Ct is defined as the concentration at specified time "t".
Correlation Between Ct and/ or AUC versus the Change in Plasma HIV-1 RNA (Log10 Copies/mL) from Day 1 Through Day 11 | Day 1 up to Day 11
Percentage of Participants at Any Measurement Achieving HIV-1 RNA < 50 Copies/mL by Day 11 at Each Dose Level | Up to Day 11
Percentage of Participants With Emergence of Viral Resistance to the ARV Class of the Given Drug (GS-1219) | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (15):
- United States (15):
  - Ruane Clinical Research Group, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Washington Health Institute, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, DeLand, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - BLISS Health Inc, Orlando, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute, West Palm Beach, Florida
  - Be Well Medical Center, Berkley, Michigan
  - Central Texas Clinical Research, Austin, Texas
  - Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - AXCES Research Group, El Paso, Texas
  - AXCES Research Group, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT07115368